CLINICAL TRIAL: NCT02411643
Title: Molecular Effects of Topical Calcipotriene on Morphea
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Accrual incomplete/Investigator left institution
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Lauren Graham, Clinical Instructor in Dermatology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00101294
Record Dates: First submitted 2015-03-03; First posted 2015-04-08 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2017-12

CONDITIONS: Morphea; Localized Scleroderma
MeSH Terms: conditions — Scleroderma, Localized | interventions — calcipotriene; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- topical calcipotriene 0.005% ointment (Other): Calcipotriene 0.005% applied to affected areas twice daily to all enrolled subjects
  Interventions: Drug: topical calcipotriene 0.005% ointment

INTERVENTIONS:
Drug: topical calcipotriene 0.005% ointment — Affected area will be treated twice daily for 3 months
  Other Names: Dovonex

SUMMARY:
This study will look into how topical treatment with synthetic Vitamin D3, calcipotriene ointment, used as standard of care, works in patients with morphea. Skin biopsies of morphea lesions before and after treatment with topical calcipotriene 0.005% ointment will be analyzed for changes in RNA and protein. A skin biopsy of unaffected skin will also be obtained and used for a control. This is an initial study to look at the molecular effects of topical calcipotriene on human morphea-involved skin. This study will look at the differences between affected and unaffected skin. This study also will look at clinical outcomes in morphea patients and determine if there are any clinical predictors for improvement with the medication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinically-diagnosed or biopsy proven plaque-type, guttate, linear, segmental, and generalized morphea that are receiving calcipotriene 0.005% ointment as part of their standard of care treatment will be included.
* Subjects are allowed to have previously been on any therapy as long as they have been off systemic treatment, topical therapy or phototherapy for 4 weeks prior to baseline.
* Age ≥ 18 years.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Subjects with the diagnosis of morphea profundus, eosinophilic fasciitis, and atrophoderma will be excluded.
* Subjects who are receiving oral or topical immunosuppression therapy or phototherapy within 4 weeks prior to entering the study.
* Subjects may not be receiving any investigational agents.
* Subjects must not be pregnant or nursing.
* Patients allergic to lidocaine or epinephrine or who have a history of impaired wound healing or for any reason are unable to undergo a skin biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topical Calcipotriene 0.005% Ointment
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Topical Calcipotriene 0.005% Ointment
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change of Gene Expression From Skin Biopsy
Description: Skin biopsy will be taken at day 0 and 3 months, RNA will be looked at for different gene expression levels
Time Frame: day 0 and 3 months
Population: Study was terminated prior to obtaining results.
Arm/Group | Topical Calcipotriene 0.005% Ointment
Number analyzed (Participants) | 0

2. Secondary Outcome: Quality of Life
Description: Quality of life questions will be asked at day 0 and 3 months
Time Frame: day 0 and 3 months
Population: Study was terminated prior to obtaining results.
Arm/Group | Topical Calcipotriene 0.005% Ointment
Number analyzed (Participants) | 0

3. Secondary Outcome: Modified Localized Scleroderma Skin Score
Description: The firmness or tightness of the skin will be measured throughout the body at day 0 and 3 months
Time Frame: day 0 and 3 months
Population: Study was terminated before results were obtained.
Arm/Group | Topical Calcipotriene 0.005% Ointment
Number analyzed (Participants) | 0

4. Secondary Outcome: Change of Appearance of Skin Biopsy
Description: Skin biopsy will be taken at baseline and 3 months, skin will be examined for expression levels of different proteins
Time Frame: day 0 and 3 months
Population: Study was terminated before results were obtained.
Arm/Group | Topical Calcipotriene 0.005% Ointment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Topical Calcipotriene 0.005% Ointment
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No